CLINICAL TRIAL: NCT02913001
Title: The Effect of a Low Glycemic Load Diet on Hormonal Markers Associated With Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Nutrisystem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: New York University
Record Dates: First submitted 2016-09-03; First posted 2016-09-23 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2016-09

CONDITIONS: Acne Vulgaris
Keywords: Diet; glycemic index; glycemic load; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Glycemic Load Diet (Experimental): Participants received a diet education to follow a low glycemic load diet and received some low glycemic load staple foods.
  Interventions: Other: Low Glycemic Load Diet
- Usual Eating Plan (Active Comparator): Participants received a diet education to continue with their usual diet.
  Interventions: Other: Usual Eating Plan

INTERVENTIONS:
Other: Low Glycemic Load Diet — Participants received a diet education on a low glycemic load diet.
  Arms: Low Glycemic Load Diet
Other: Usual Eating Plan — Participants received a diet education to continue with their usual eating plan.
  Arms: Usual Eating Plan

SUMMARY:
This randomized controlled trial will examine changes in some hormonal markers associated with acne among adults with moderate/severe acne randomized to a low glycemic index and glycemic load diet or usual eating plan for two weeks.

DETAILED DESCRIPTION:
The objectives of this randomized controlled trial are to investigate the impact of a low glycemic index/load eating plan on endocrine aspects of acne. Specifically, this study will examine changes in blood biochemical markers of acne among adults with acne following a modified carbohydrate (low glycemic index/load) eating plan or their usual eating plan for two weeks. An external sponsor, Nutrisystem®, will provide some low glycemic index/load foods to the study participants randomized to the intervention group for two weeks. Study outcomes include changes in glucose, insulin, insulin resistance, insulin-like growth factor-1, and insulin-like growth factor binding protein-3 concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 or <30.0 kg/m2
* History of moderate or severe facial acne for at least 6 months
* Able to read and speak the English language

Exclusion Criteria:

* > 10% weight change within the last 6 months
* Taking medications known to alter blood glucose or insulin concentrations
* Medical history of polycystic ovarian syndrome, type 1 diabetes, type 2 diabetes, or pre diabetes
* Low carbohydrate (<45% of total energy from carbohydrate), glycemic index, or glycemic load diet
* Female participants that are pregnant or lactating or were pregnant or lactating within the last year
* Current use of a pacemaker or other battery operated implant
* Facial hair that would make it difficult for a health care provider to assess facial acne.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
blood glucose in mg/dL | Change from baseline blood glucose concentrations after two weeks.
  A trained clinician will use venipuncture to draw approximately 30 mL of blood to measure glucose concentrations
Insulin in uIL/mL | Change from baseline insulin concentrations after two weeks.
  A trained clinician will use venipuncture to draw approximately 30 mL of blood to measure insulin concentrations
Insulin-like growth factor-1 in ng/mL | Change from baseline Insulin-like growth factor-1 concentrations after two weeks.
  A trained clinician will use venipuncture to draw approximately 30 mL of blood to measure insulin-like growth factor-1 concentrations
Insulin-like growth factor binding protein-3 in mg/L | Change from baseline insulin-like growth factor binding protein-3 concentrations after two weeks.
  A trained clinician will use venipuncture to draw approximately 30 mL of blood to measure insulin-like growth factor binding protein-3 concentrations

SECONDARY OUTCOMES:
Changes in Acne specific quality of life among participants following a low glycemic load diet or their usual diet for two weeks. | Change in baseline quality of life after two weeks.
  Acne specific quality of life will be measured using a validated questionnaire. Acne specific quality of life measured the effect of acne on the participants quality of life.

OTHER OUTCOMES:
Changes in nutrition self efficacy among participants following a low glycemic load diet or their usual diet for two weeks | Change in nutrition self-efficacy after two-weeks.
  Nutrition self-efficacy, or the ability to make diet changes, will be measured using a validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Woolf, PhD, Principal Investigator — New York University; Jennifer Burris, PhD, Study Director — New York University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burris J, Rietkerk W, Woolf K. Acne: the role of medical nutrition therapy. J Acad Nutr Diet. 2013 Mar;113(3):416-430. doi: 10.1016/j.jand.2012.11.016. PMID 23438493
- [Derived] Burris J, Shikany JM, Rietkerk W, Woolf K. A Low Glycemic Index and Glycemic Load Diet Decreases Insulin-like Growth Factor-1 among Adults with Moderate and Severe Acne: A Short-Duration, 2-Week Randomized Controlled Trial. J Acad Nutr Diet. 2018 Oct;118(10):1874-1885. doi: 10.1016/j.jand.2018.02.009. Epub 2018 Apr 22. PMID 29691143